CLINICAL TRIAL: NCT03635723
Title: Breast: Recovery After Axillary Node Clearance - Evaluating Limbs With E-Technology (the BRACELET Study)
Acronym: BRACELET
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/LO/1038 BRACELET
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Mobility Limitation
Keywords: Technology; Rehabilitation; Wearables; Breast surgery; Physical activity; Enhanced recovery after surgery
MeSH Terms: conditions — Breast Neoplasms; Mobility Limitation; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgical: Having undergone a procedure in hospital
  Interventions: Device: Activity monitor

INTERVENTIONS:
Device: Activity monitor — Technology allowing measurement of physical activity

SUMMARY:
This work aims to use wearable sensors to record the return towards normal physical activity after breast surgery. It will build on current evidence by using objective measures of activity and arm movements rather than patient reports.

ELIGIBILITY:
Inclusion Criteria:

* Breast or axillary surgery

Exclusion Criteria:

* Other diagnosed movement disorder
* Cannot consent due to language or capacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Arm movements | Post-operative for 2-4 weeks
  Arm movements as measured by wearable sensor

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kwasnicki, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom